CLINICAL TRIAL: NCT02682017
Title: Effect of Consuming Pork From Animals Supplemented With Laminarin and Fucoidan Derived From the Brown Seaweed Laminaria Digitata on the Antioxidant Status of Human Participants.
Brief Title: Effect of Consuming Pork From Seaweed Extract Fed Animals on Antioxidant Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University College Dublin (Other); University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REC/11/0080
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Antioxidant Status, Inflammation
Keywords: Seaweed; Pork; Fucoidan; Laminarin; Functional Food; Antioxidant activity
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Placebo Comparator): Pork meat from pigs feed with a standard feed
  Interventions: Other: Pork meat from pigs feed with a standard feed.
- Treatment 2 (Experimental): Pork meat from pigs fed a feed with a Laminarin/fucoidan mix
  Interventions: Other: Pork meat from pigs fed a feed with a Laminarin/fucoidan mix

INTERVENTIONS:
Other: Pork meat from pigs feed with a standard feed. — 4 week intervention with 700g (raw weight) of pork meat (3x pork burgers (125g raw weight each) + pork mince (325 g raw weight) per week.
  Arms: Treatment 1
Other: Pork meat from pigs fed a feed with a Laminarin/fucoidan mix — 4 week intervention with 700g (raw weight) of pork meat (3x pork burgers (125g raw weight each) + pork mince (325 g raw weight) per week from pigs fed animal feed supplemented (5.37 kg/tonne of feed) with spray-dried laminarin and fucoidan (seaweed).
  Arms: Treatment 2

SUMMARY:
Red meat makes a significant contribution to the human diet. The most widely consumed meat globally is pork which accounts for 36% of overall meat intake with beef and poultry contributing 22% and 35%, respectively. Pork meat provides a range of important nutrients including protein, zinc, B-vitamins and a range of important minerals however there is accumulating evidence to suggest that consuming red meat and processed meat increases the risk of cardiovascular disease (CVD) and colon cancer. Despite these reports of a negative impact on health, global pork consumption continues to increase and there are increasing efforts to improve the nutritional profile of pork meat through the development of novel porcine feed regimens. The manipulation of pig feed to produce 'healthier' meat and meat products offers a feasible approach to reduce the risk of preventable disease. Furthermore, recent projections of an increased global demand for pork and poultry, particularly in China, have highlighted the increasing strain that will be placed on the supply of grains and the need to find alternative and sustainable feed ingredients. Macroalgae is emerging as a potential sustainable source of novel bioactive ingredients for the animal feed industry with some species known to be a good source of protein, minerals, polyunsaturated fatty acids and a range of fibre components including fucoidan and laminarin.

The polysaccharides, laminarin and fucoidan, which are found in abundance in brown seaweed, are gaining increasing attention as a potential bioactive feed ingredients with putative antioxidant, anti-inflammatory and immunomodulatory activities. Incorporation of a laminarin/fucioidan mix (LAM/FUC) into the porcine diet was shown to result in lower levels of lipid oxidation in fresh pork steaks. Numerous studies to date have also investigated the health promoting effects of LAM/FUC through modulation of the porcine gut microbiota which was shown to enhance inflammatory cytokine expression in response to pathogen recognition and also to increase piglet performance post weaning.

The uptake and fate of fucoidan in humans remains unknown albeit after consumption, unaltered fucoidan has been detected in human plasma after ingestion suggesting at least partial bioavailability of this compound. A study by Moroney et al. (2015) using an in vitro bioavailability Caco-2 model provided indications that fucoidan was bioavailable and that it may have potent antioxidant potential.

The primary aim of this randomised parallel placebo controlled human intervention trial was to investigate if consuming pork meat from pigs supplemented with a LAM/FUC mix, in addition to their normal diet, would impact on blood oxidant and inflammatory status of healthy adults. The secondary aim was to determine the effect of consuming LAM/FUC fed pork meat on lymphocyte DNA damage, lipid status and immune function in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-55 years
* Non smoking
* BMI of < 18.5 or > 30 kg/m2.

Exclusion Criteria:

* Regular consumers of seaweed (>5 g/week)
* Non-consumers of pork or pork products
* Smoker
* Pregnant and lactating women
* Vegetarians and vegans
* Lactose intolerant individuals
* Diabetes
* Cardiovascular disease
* Autoimmune/ inflammatory disorders
* History of neoplasm
* Recent acute illness and/or chronic prescribed or self-prescribed use of anti-inflammatory agents (including aspirin)
* Use of broad spectrum antibiotics
* Use of drugs active on gastrointestinal motility or laxatives
* Use of dietary supplements (specifically probiotics or prebiotics).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in antioxidant status | Baseline + 4 weeks
  Plasma Ferric Reducing Antioxidant Power

SECONDARY OUTCOMES:
Change in protection against DNA damage | Baseline + 4 weeks
  Lymphocyte DNA damage prior to and following an oxidative challenge with hydrogen peroxide.
Change in serum lipid profile | Baseline + 4 weeks
Change in plasma inflammatory status | Baseline + 4 weeks
  C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom